CLINICAL TRIAL: NCT03661580
Title: Integrating Behavioural Activation for Depression Into Community Drugs and Alcohol Treatment: A Randomised Controlled Trial
Brief Title: BA Trial for Co-Occurring Depression and Substance Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Sophie Pott, PhD Student, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URMS: 157527
Record Dates: First submitted 2018-09-04; First posted 2018-09-07 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Depression; Substance Use Disorders
MeSH Terms: conditions — Depression; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This study is a pragmatic, parallel group, randomised controlled trial assessing the efficacy of BA compared to treatment as usual (TAU) for patients with depression who are accessing Community Drugs and Alcohol Treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioural Activation (Experimental): Participants in this arm receive 6 x weekly 1:1 sessions of BA delivered by a trained drugs and alcohol worker at the CDAT service. At the end of the 6-week intervention period participants will be referred back to their usual caseworker at the CDAT service, though they will be offered two BA booster sessions with their BA worker at 2-3 weeks and 4-5 weeks post-treatment. All participants in this arm will continue to have access to Treatment as Usual (i.e. prescribing) as required throughout the intervention period.
  Interventions: Behavioral: Behavioural Activation
- Treatment as Usual (Active Comparator): Participants in this arm will receive no change to the care they usually receive at the CDAT service.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Behavioural Activation — The BA intervention will be the outpatient version of the Life Enhancement Treatment for Substance Use (LETS ACT; Daughters et al., 2008). This brief, manualised BA intervention has been specifically developed to meet the needs of patients with comorbid substance misuse and depression in drugs and alcohol treatment settings. LETS ACT targets the link between mood, substance use and behaviour, and focuses on identifying and increasing rewarding, substance-free activities that are based on the patient's own personal values.
  Other Names: LETS ACT
  Arms: Behavioural Activation
Behavioral: Treatment as Usual — The control intervention in this study is Treatment as Usual at the CDAT service. Treatment as Usual consists of planned key-working sessions every 2-4 weeks with an allocated caseworker plus monthly prescribing review appointments with a medical practitioner for patients who require drug treatment medication. Key-working sessions are primarily focused on addressing substance misuse issues using a range of intervention techniques such as motivational interviewing and brief solution-focused therapy.
  Arms: Treatment as Usual

SUMMARY:
A large proportion of people seeking treatment for drug and alcohol issues also have clinically significant depression symptoms. This combination of problems tends to have a negative impact on treatment and leads to poor health and disability, yet relatively few studies have focused on the development of interventions for treating this comorbidity. There is emerging evidence to suggest that Behavioural Activation (BA) may be a viable and cost-effective treatment for comorbid depression and substance use problems, however more research is needed in order to establish its effectiveness in routine practice. The aim of this study is therefore to investigate the efficacy of a brief (6-session), manualised BA intervention among service users with depression who are accessing Community Drugs and Alcohol treatment. We are planning to recruit up to 128 service users who are actively using substances to be randomly assigned to either the 6-week BA intervention or Treatment as Usual in Community Drugs and Alcohol services. These participants will be recruited from either a Community Drugs and Alcohol service or a Community Mental Health service. Our research will assess whether the BA intervention is more effective than usual care in (1) reducing depression symptoms, (2) reducing substance use, and (3) improving treatment engagement (i.e. session attendance). We expect that our results will establish the efficacy of integrating BA for depression into routine Community Drugs and Alcohol Treatment.

DETAILED DESCRIPTION:
RATIONALE Over 50% of treatment-seeking substance users present with clinically significant depression symptoms (Johnson, Neal, Brems, & Fisher, 2006). This combination of problems tends to complicate treatment (e.g. Carroll et al., 1993) resulting in greater functional impairment (Johnson et al., 1995) and poor health outcomes (Hasin et al., 2002). Treatment protocols for co-occurring mental health and substance misuse have traditionally focused on treating these issues separately, however there is now increasing consensus that integrated approaches to treatment are more effective (Davidson et al., 2010) and subsequently a growing interest into how targeted mental health support can be incorporated into standard drug and alcohol treatment.

CBT is deemed to be one of the most effective psychological treatments for depression, though may be too complex and time-consuming for effective delivery in routine CDAT. Emerging evidence suggests that a more suitable intervention in this context may be Behavioural Activation (BA); a brief, manualised intervention which targets depression symptoms by increasing engagement in rewarding, values-based activities (Lejuez, Hopko, Acierno, Daughters, & Pagoto, 2011). Indeed, previous studies have found that BA is associated with reductions in both depression symptoms and substance use (Daughters et al., 2018; Daughters et al., 2008; Delgadillo et al., 2015), as well as improved treatment retention among substance misuse service users with comorbid depression (Magidson et al., 2011). The only known trial of BA in UK Community Drugs and Alcohol Treatment (CDAT) was conducted by Delgadillo and colleagues (2015), however this study was under-powered and employed qualified mental health practitioners to deliver the intervention which may be too costly or unfeasible to implement in routine practice. More research is needed to establish the efficacy of BA in CDAT services, and given that BA may be delivered effectively with minimal training by staff who are not formally trained as psychological therapists (Ekers et al., 2008), it seems that the most suitable and cost-effective way of integrating BA into routine drug and alcohol treatment would be to upskill the existing workforce.

Accordingly, given the high prevalence and impact of comorbid depression among addiction service users, along with evidence to suggest that BA is an effective and acceptable intervention for treating this population, the present study will expand on previous research by conducting a trial to evaluate the efficacy of BA delivered by trained drugs and alcohol workers in a sample of patients accessing treatment for substance use. The central research question is: How effective is Behavioural Activation for treating depression in substance users compared to treatment as usual in Community Drugs and Alcohol services?

AIMS

The proposed study aims to:

1. Evaluate the efficacy of brief one-to-one manualised BA delivered by trained drugs and alcohol workers in a CDAT setting in terms of depression outcome
2. Evaluate the efficacy of delivering manualised BA in this setting in terms of substance use and engagement (attendance and dropout rates) outcomes

HYPOTHESES

Participants who receive the BA intervention will show improvements in:

1. Depression symptoms
2. Substance use
3. Treatment Engagement (sessions attended, % dropout)

CLINICAL IMPLICATIONS If the BA intervention is found to be more effective than the usual care offered in CDAT services, this trial will provide evidence for the intervention to be implemented in routine practice. Even if the BA intervention is not found to be more effective, the results of this study will contribute to understanding of what works and what doesn't work in this setting, which can be used to inform the development of future interventions aimed at addressing co-occurring substance use and depression.

DESIGN This study is a pragmatic, parallel group, randomised controlled trial assessing the efficacy of BA compared to treatment as usual (TAU) for patients with depression who are accessing CDAT services. Outcome measures will be taken at baseline, 3-, 6-, 12- and 24-weeks to enable the comparison of relative efficacy.

METHOD Participants will be recruited from CDAT services in the UK. They will be working age adults (18-65) with mild to moderate depression who are actively using substances. The study aims to recruit 142 participants in total.

PROCEDURE Drugs and alcohol workers in CDAT services will employ a step-wise mental health screening strategy as part of routine practice in order to identify potential participants. This strategy involves routinely completing TOP and brief mental health questionnaires sequentially in order to identify patients with common mental disorders.

Potential participants will be provided with an information sheet and asked for permission to pass their details on to the research team.

Consenting participants will be contacted by a member of the research team within one week to conduct eligibility screening and obtain informed consent. Participants will be aware of confidentiality arrangements for the study, that their participation is voluntary and that they have the right to withdraw at any time.

Once consent to participate has been established, the identified clients' details will be passed on to an independent administrator for randomisation.

Participants will be randomly allocated into one of two arms ('BA Intervention' or 'Treatment as Usual'). Participants randomised to Treatment as Usual will continue to receive their usual care at the CDAT service. Participants randomised to the BA intervention will receive 6 x weekly one-to-one sessions of BA plus 2 booster sessions at 2-3 and 4-5 weeks post-treatment. BA will be delivered by drugs and alcohol workers who have completed 2 days of training in delivering the BA intervention. Staff delivering the intervention will also receive an extra hour of supervision once per month with a supervisor-trained supervisor which will be focused on delivery of the BA intervention.

To ensure fidelity to the BA treatment protocol, drugs and alcohol workers delivering the BA intervention will complete a checklist at the end of each session indicating their adherence to the session protocol, with the checklist for each session highlighting specific session objectives. Additionally, drugs and alcohol workers will be asked to audiotape at least two of their sessions at random over the course of the study. Audiotaped therapy sessions will be rated using the rating scales from Magidson and colleagues' (2011) study by an independent evaluator with an understanding of behavioural activation strategies. Independent evaluators will be Psychological Wellbeing Practitioners with experience of delivering BA, the Study Coordinator, or students under the supervision of the Study Coordinator. Issues of non-adherence will be considered a training implication representative of areas for improvement to be addressed via standard supervisory procedures. Non-adherence will not preclude data inclusion for the purposes of this study; instead it will be addressed as a limitation of the study related to therapist experience.

DATA ANALYSIS Screening, recruitment, random allocation and treatment engagement (including dropout) data will be summarised using a CONSORT diagram. The integrity of randomisation, demographic and clinical characteristics will be assessed by comparing between groups and between recruitment sites using appropriate statistical tests. Loss to follow-up has been estimated at 20% based on a previous feasibility study of BA conducted in this setting (Delgadillo et al., 2015). Intention-to-treat analyses will be conducted using Last Observation Carried Forward method in order to account for the loss to follow-up. Secondary to this, we will analyse the data only with participants who completed all of the follow-up assessments in order to check that findings were not unduly affected by attrition.

We will calculate and report standardised effect sizes for depression outcome (PHQ-9) using Cohen's d. Severity of depression at 12-week follow-up will be considered the main outcome for the calculation of effect sizes; although we will also report 6- and 24-week follow up data for comparison. Severity of depression at 12-week follow-up will be compared between-groups using Analysis of Covariance with participant's pre-treatment scores on the PHQ-9 used as covariates. This is to counter potential baseline variance in depression that may influence results and was considered robust for relatively small sample sizes in a similar study of BA (Ekers et al., 2011).

For both intervention and control groups, we will present the proportions of participants who had reliable and clinically significant change (RCSC) in depression status at 6, 12 and 24 weeks. The RCSC outcome definition (Jacobson & Truax, 1991) has been recommended as a standard reporting strategy for all published research involving psychological interventions (Evans et al., 1998).

Pre-post changes scores will also be calculated and reported for substance use outcomes (Percent Days Abstinent and Severity of Dependence). Percent days abstinent will be considered the primary substance use outcome. We will calculate and report standardised effect sizes for percent days abstinent at 12-week follow-up using Cohen's d, with 6- and 24-week follow-up data reported for comparison. Percent days abstinent at 12-week follow-up will then be compared between groups using Analysis of Covariance, with participant's pre-treatment scores on the SDS entered as a covariate to account for potential baseline variance in severity of dependence that may influence results. Changes in SDS scores pre-post treatment will be compared between groups using Student's t-test.

For both intervention and control groups, we will present the proportions of participants who had reliable and clinically significant change (RCSC) in percent days abstinent and severity of dependence at 6, 12 and 24 weeks based on guidelines by Jacobson and Truax (1991).

The mean number of key-working sessions offered to participants in the Treatment as Usual arm during the 6-week intervention period will be reported. Percentage of sessions attended will then be compared between groups using Student's t-test.

SAMPLE SIZE CALCULATION Based on previous research conducted in the USA, an effect size of 0.5 was used to calculate the required sample size (Daughters et al., 2018; Daughters et al., 2008). Standard sample size calculation based on a medium effect size (0.5) with 2 independent sample means indicates that 128 participants (64 per group) would be required to achieve 80% power using a significance level (p) of 0.05. After accounting for the possibility that an estimated 10% of participants may drop out of the study (i.e. withdraw consent), this means that we will need to recruit 142 participants in total (71 per group). A previous feasibility study conducted by Delgadillo and colleagues (2015) indicated a screened to recruited ratio of 4:1 in this setting, therefore we will aim to screen a minimum of 568 participants sequentially over a 2-year period in order to achieve an adequate sample size for this study.

ELIGIBILITY:
Inclusion Criteria:

* Are currently engaging with a Community Drugs and Alcohol Treatment (CDAT) service. Engagement is defined by (a) being currently registered with the service and (b) having had planned contact with the service within the last month.
* Meet criteria for a current depressive disorder as defined by a score of 12 or more on the PHQ-9 questionnaire. Comorbid anxiety disorders are not exclusion criteria, as long as depression is the primary disorder.
* Meet criteria for mild-to-moderate severity of drug dependence, as defined by a score between 0 - 10 on the Severity of Dependence Questionnaire.
* Have used alcohol or illicit drugs within the last month.

Exclusion Criteria:

* Are not currently engaging with a Community Drugs and Alcohol Treatment (CDAT) service
* Are assessed as having a high risk of suicide warranting involvement with crisis services
* Have an organic or acquired brain injury
* Do not currently meet criteria for depressive disorder as defined by the PHQ-9 questionnaire score.
* Meet criteria for depression and a comorbid anxiety disorder, as identified by the GAD-7 questionnaire. Where the anxiety disorder is more severe, has been of longer duration than depressive symptoms and is the patient's main concern.
* Patients with severe mental health problems who are already involved in psychiatric or secondary care mental health services.
* Are free of substances of dependence
* Those who have a severe drug or alcohol dependence, as defined by a score above 10 on the Severity of Dependence Questionnaire.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 12 weeks
  Change in depression at post-treatment follow-up via the PHQ-9 (Kroenke et al., 2001). The PHQ-9 is a brief (9-item) self-report 4-point Likert-type scale measure is based on the Diagnostic and Statistical Manual (DSM-IV) diagnostic criteria for major depressive disorder. Each item is rated on a 0 to 3 scale relating to the frequency of depressive symptoms over the last two weeks (0 = 'not at all', 3 = 'nearly every day'). Scores range from 0 to 27 with higher scores indicating a greater severity of depression.

SECONDARY OUTCOMES:
Percent Days Abstinent | 12 weeks
  Change in Percent Days Abstinent at post-treatment follow-up via the Treatment Outcomes Profile (TOP)
Severity of Dependence | 12 weeks
  Change in Severity of Dependence to the primary drug at post-treatment follow-up via the Severity of Dependence Scale (SDS; Gossop et al., 1995). The SDS is a brief (5-item) self-report 4-point Likert-type scale measure used to assess the severity of dependence to a drug. Scores range from 0 - 15, with higher scores indicating greater psychological dependence.

OTHER OUTCOMES:
Treatment Engagement | 6 weeks
  Difference in percentage of treatment sessions attended between participants allocated to BA and Treatment as Usual

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Delgadillo, Study Director — University of Sheffield
Locations (1):
- Aspire Drug and Alcohol Service, Doncaster, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No